CLINICAL TRIAL: NCT01760538
Title: Study on Heart Rate Variability in Cardiac Transplant Recipients With Exercise and After Exercise Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1913; NSC 90-2314-B-002-313; NSC 91-2314-B-002-320
Record Dates: First submitted 2013-01-02; First posted 2013-01-04 (Estimated); Last update posted 2013-01-04 (Estimated); Status verified 2012-11

CONDITIONS: Cardiac Transplant Disorder
Keywords: Cardiac transplant recipients; Heart rate variability; Exercise training
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- exercise group (Experimental): exercise training
  Interventions: Behavioral: Exercise training
- Control (Active Comparator): usual care
  Interventions: Behavioral: usual care

INTERVENTIONS:
Behavioral: Exercise training — exercise training
  Arms: exercise group
Behavioral: usual care — received usual medical care after heart transplantation
  Arms: Control

SUMMARY:
The purpose of the study was to investigate the changes on heart rate variability, exercise capacity, activities of daily living, and quality of life after aerobic exercise training in cardiac transplant recipients.

ELIGIBILITY:
Inclusion Criteria:

* Heart transplant recipients with stable post operation condition
* Age between 20-70 years
* No acute or severe chronic rejection

Exclusion Criteria:

* Any condition that might affect exercise performance

Ages: 20 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2001-08; Primary Completion 2003-09 (Actual); Study Completion 2003-09 (Actual)

PRIMARY OUTCOMES:
Heart rate variability | 8 weeks
  R-R interval difference

SECONDARY OUTCOMES:
Exercise capacity | 8 weeks
  oxygen consumption
Quality of life | 8 weeks
  This outcome measures how good life the patients have

CONTACTS AND LOCATIONS:
Overall Officials: Ying-Tai Wu, Doctor, Study Director — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan